CLINICAL TRIAL: NCT05363891
Title: Phase II, Double-blind, Placebo-Controlled, Randomized Trial Examining Natrunix in Combination With Methotrexate (+Folate) for the Treatment of Rheumatoid Arthritis
Brief Title: Natrunix or Placebo in Combination With Methotrexate in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XBiotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-PT055
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Arm 1- Natrunix 200mg with MTX(+Folate) Arm 2 - Natrunix 400mg with MTX(+Folate) Arm 3- Placebo with MTX(+Folate)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Natrunix 200mg with MTX(+Folate) (Experimental): Natrunix 200mg, subcutaneous injection in combination with Methotrexate (+Folate).This arm will enroll 70 subjects.
  Interventions: Drug: Natrunix
- Natrunix 400mg with MTX(+Folate) (Experimental): Natrunix 400mg, subcutaneous injection in combination with Methotrexate (+Folate).This arm will enroll 70 subjects.
  Interventions: Drug: Natrunix
- Placebo with MTX(+Folate) (Placebo Comparator): Placebo in combination with Methotrexate (+Folate).This arm will enroll 70 subjects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Natrunix — Natrunix is a unique kind of drug-an immunoglobulin cloned from a naturally occurring immune response from a healthy human donor. Natrunix blocks inflammation in a unique way-it is the only therapeutic that exclusively neutralizes interleukin-1α (IL-1α), a crucial mediator of interleukin-1 inflammation. Targeting IL-1α directly using a natural human monoclonal antibody may provide a safer and more effective means of blocking interleukin-1 in rheumatoid arthritis.
  Other Names: True Human IgG4 monoclonal antibody
  Arms: Natrunix 200mg with MTX(+Folate); Natrunix 400mg with MTX(+Folate)
Drug: Placebo — Placebo
  Arms: Placebo with MTX(+Folate)

SUMMARY:
Phase II, Double-Blind, Placebo-Controlled, Randomized Trial Examining Natrunix in Combination with MTX (+Folate) for the Treatment of Rheumatoid Arthritis

DETAILED DESCRIPTION:
Potential subjects will be consented and screened for study eligibility and the enrolled will be randomized in a 1:1:1 ratio to receive either: 200 mg Natrunix; 400mg Natrunix; or placebo. All subjects will enter the study on stable MTX dose. Subjects will receive once weekly injection of Natrunix or placebo in addition to MTX for 12 weeks. The study will conclude after 13 weeks.

Study Duration is 17 weeks (4-week maximum screening + 12-week treatment period = 1-week follow-up.

The primary objective is to determine the ACR 20 response rate in subjects receiving stable dose of MTX and after 12 weeks of treatment with either Natrunix or placebo. The study will also examine what impact the addition of Natrunix or placebo has on the scores of various rheumatological grading scales, including ACR 50, NRS-pain score, and 66/68-joint count, as well as safety. All subjects enrolled in the study will be taking concomitant methotrexate.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study if they meet all of the following criteria:

1. Weight > 40 kg
2. Diagnosis of moderate to severe RA according to 2010 ACR/EULAR classification criteria.
3. Patients must be methotrexate-inadequate responders.

   a. Persistent moderate to severe RA disease activity (ie. criteria #2 above) despite ongoing treatment with MTX.
4. Meets the following minimum disease activity criteria at screening: ≥6 swollen joints (based on DAS28) and ≥6 tender joints (based on DAS28) and DAS-ESR > 3.2.
5. Subject must be receiving MTX treatment at a dosage of 15-25 mg/week for a minimum of12 weeks; and be receiving a stable dose of MTX for >4 weeks preceding randomization.

   Subjects must also be in principle agreement to remain at the pre-randomization stable dose of MTX for the entire duration of the study. Subjects must also be willing to take a minimum of 5 mg folic acid/folinic acid per week for the duration of the study.
6. Male or female, at least 18 years of age, willing to provide informed consent, able to attend all clinic visits,comply with study-related procedures and able to understand and complete study-related questionnaires.
7. Patients must provide at least 7 consecutive days of NRS-pain data in the subjects diary prior to the baseline visit. The NRS pain diary should ideally be completed for the 7 days immediately prior to Visit 1 (when the first dose of test drug is administered). Subjects may record more than 7 days of pain records in the diary for their baseline. At least seven consecutive days of pain diary are necessary to be eligible for enrollment in the study.
8. Peripheral blood CD19+ cell count recovery to >10 cells/uL or >1% of total lymphocyte count (Required only for subjects who have received a Rituximab (or anti-CD20 biosimilar) infusion within 12 months prior to enrollment).
9. Female patients of childbearing potential must consent to undergo a serum pregnancy test at enrollment, and urine pregnancy tests at each visit after screening. Women of non-childbearing potential include those considered to have a medical history that indicates that pregnancy is not a reasonable risk, including post-menopausal women and those with a history of hysterectomy or surgically sterilized.
10. In case of female patients of childbearing potential, willingness to use one method of contraception of high efficacy during the entire study period. These methods can include but not limited to hormonal contraceptives, intrauterine devices, condoms, diaphragms, etc.
11. Males participating in this clinical research study should not get a sexual partner pregnant during their participation in this research study as the effect of the study drug on sperm is not known. Male contraception methods can include but are not limited to mechanical methods (e.g., abstinence, non-vaginal intercourse), contemporary methods comprising barrier methods (e.g., spermicide, condom, sponge, diaphragm and cervical cap) and vasectomy.

Exclusion Criteria:

Patients with ANY of the following will be excluded from the study:

1. History of treatment with Natrunix for any reason.
2. Any active, chronic, or recurrent infections. (e.g., ongoing bacterial, viral, or fungal infection).
3. Comorbid severe psychiatric illness and/or complicated social situations that would limit compliance with study requirements.
4. Patients with a positive result of TB test (QuantiFERON-TB Gold (QFT) at screening unless the patients can present a documentation of completion of TB treatment course by the local Health Department and a clear chest x-ray at enrollment.
5. Patients must not have received any biological therapy including anakinra, rilonacept, canakinumab, adalimumab, certolizumab, etanercept, golimumab, infliximab, abatacept, tocilizumab, sarilumab, and biosimilars within 8 weeks prior to randomization.
6. Treatment with JAK inhibitors within 4 weeks (or 5 half-lives, whichever is longer) prior to randomization.
7. Investigational therapy administered within a time interval less than at least 5 half-lives of the investigational agent prior to the first scheduled day of dosing in this study.
8. Pregnant or breastfeeding patients.
9. Patients with current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within a year prior to Day 0.
10. Uncontrolled heart disease, including NYHA Class III or IV congestive heart failure, ventricular arrhythmia, uncontrolled blood pressure (defined as ≥ 160/100 mm Hg), or unstable angina.
11. Clinically significant laboratory abnormalities, including:

    1. Hemoglobin <9.0 g/dL
    2. White blood cell counts < 4000/mm3
    3. Absolute neutrophil count (ANC) <1500/mm3
    4. Platelet count <100,000/mm3
    5. Absolute lymphocyte count (ALC) <500/mm3
    6. eGFR <60 mL/min
    7. Alanine Aminotransferase (ALT) >1.5x lab upper limit of normal (ULN)
    8. Aspartate Aminotransferase (AST) >1.5x lab upper limit of normal (ULN)
    9. Bilirubin >1.5x lab upper limit of normal (ULN)
    10. GGT: Natrunix does not put any load on the liver. GGT levels are not assessed to determine potential risk of hepatoxicity. Rather GGT levels are used as an additional screening measure to assess for occult hepatobiliary disease that may be missed with more common liver enzyme assays given the requirement for concurrent treatment with therapeutic methotrexate throughout the study. Small excursions from normal values are acceptable based on Physician/Sponsor judgment.
12. Major surgery (including joint surgery) within 3 months of baseline.
13. Patients who have suffered severe trauma or fracture within 4 weeks of baseline.
14. Evidence of active hepatitis B, hepatitis C, or HIV infection.

    1. Patients positive for HBsAg and/or positive for anti-HBc antibody (regardless of anti-HBs antibody status) are excluded.
    2. Patients who are positive for Hepatitis C antibody and negative when the Hepatitis C RNA-PCR assay is performed on a subsequent sample will be eligible to participate. Patients who are positive for Hepatitis C antibody and have a positive result for the HCV when the Hepatitis C RNA-PCR assay is performed on the subsequent sample will not be eligible to participate.
15. Any other concomitant disease, disorder, or condition that could interfere with the interpretation of study endpoints, or the patient's ability to participate in and complete the study., including but not limited to:

    1. Coexisting diseases which are contraindicated for MTX treatment.
    2. Cardiovascular, renal, pulmonary, gastrointestinal, or nervous system disorders that, in the opinion of the principal investigator and/or study medical monitor, make the patient not suitable for enrollment.
    3. Concurrent autoimmune disease with the exception of Sjogren's syndrome secondary to rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
ACR 20 response rate at 12 weeks. | At 12 weeks from baseline
  The ACR is a measure used in clinical practice and clinical trial to assess medication efficacy in patients with RA, by notating improvements in swelling and tenderness in designated joints, as well as improvements in at least 3 out of 5 other categories. The other categories assessed are patient global assessment of disease activity, physician global assessment of disease activity, patient reported pain scale, disability/functionality questionnaire response, and acute phase reactant levels (CRP and ESR).

SECONDARY OUTCOMES:
ACR 50 response rate at 12 weeks. | At 12 weeks from baseline
  The ACR is a measure used in clinical practice and clinical trial to assess medication efficacy in patients with RA, by notating improvements in swelling and tenderness in designated joints, as well as improvements in at least 3 out of 5 other categories. The other categories assessed are patient global assessment of disease activity, physician global assessment of disease activity, patient reported pain scale, disability/functionality questionnaire response, and acute phase reactant levels (CRP and ESR).
Mean change in NRS-pain at 12 weeks | At 12 weeks from baseline
  Numerical rating scale (NRS) is a validated measure used to assess chronic and acute pain using a 10-point rating scale. The rating for no pain is "0" and "worst possible pain" is 10.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Medvin Clinical Research, Covina, California
  - T. Joseph Raoof MD, INC, Encino, California
  - Desert Medical Advances, Rancho Mirage, California
  - Medvin Clinical Research, Riverside, California
  - Medvin Clinical Research, Tujunga, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - HARAC Research Corp, Avon Park, Florida
  - Reliable Clinical Research, LLC, Hialeah, Florida
  - Angels Clinical Research Institute, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - BioMed Research & Medical Center, LLC, Miami, Florida
  - Advanced Clinical Research of Orlando, Ocoee, Florida
  - DH Tamarac Research Center, Tamarac, Florida
  - Greater Chicago Specialty Physicians, LLC, Orland Park, Illinois
  - Greater Chicago Specialty Physicians, LLC, Schaumburg, Illinois
  - Accurate Clinical Research Inc, Lake Charles, Louisiana
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - ClinRx Research Joseph INC, Carrollton, Texas
  - Accurate Clinical Management LLC, Houston, Texas
  - Accurate Clinical Research Inc, Houston, Texas
  - Pioneer Research Solutions, INC, Houston, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Epic Medical Research, LLC, Red Oak, Texas
  - Accurate Clinical Management, LLC, Richmond, Texas
  - DM Clinical Research, Tomball, Texas
  - Overlake Arthritis and Osteoporosis Center, Bellevue, Washington